CLINICAL TRIAL: NCT00884884
Title: Aripiprazole and Topiramate on Free-Choice Alcohol Use
Acronym: AT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Robert Swift, Professor of Psychiatry and Human Behavior, National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAA-Swift-AA015753; NIH Grant 5RO1AA015753-02
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; alcohol abuse; topiramate; aripiprazole
MeSH Terms: conditions — Alcoholism | interventions — Aripiprazole; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Double Placebo (Placebo Comparator): Placebo, Placebo
  Interventions: Drug: Double Placebo
- Aripiprazole 15, Placebo (Experimental): 15 mg Aripiprazole, Placebo
  Interventions: Drug: Aripiprazole 15, placebo
- Aripiprazole 7.5, Placebo (Experimental): Aripiprazole 7.5 mg daily plus Placebo daily
  Interventions: Drug: Aripiprazole 7.5, Placebo
- Topiramate 100mg, Placebo (Experimental): Topiramate 100 mg daily plus Placebo daily
  Interventions: Drug: Topiramate 100, Placebo
- Topiramate 200, Placebo (Experimental): Topiramate 200 mg daily plus Placebo daily
  Interventions: Drug: Topiramate 200, Placebo
- Topiramate 100, Aripiprazole 5 (Experimental): Topiramate 100 daily plus, Aripiprazole 5mg daily
  Interventions: Drug: Topiramate 100, Aripiprazole 15; Drug: Topiramate 100, Aripiprazole 15mg
- Topiramate 200, Aripiprazole 15 (Experimental): Topiramate 200 mg daily plus Aripiprazole 15mg daily
  Interventions: Drug: Topiramate 200, Aripiprazole 15
- Topiramate 100, Aripiprazole 7.5 (Experimental): Topiramate 100 mg daily, Aripiprazole 7.5 mg daily
  Interventions: Drug: Topiramate 100, Aripiprazole 7.5
- Topiramate 200, Aripiprazole 7.5mg (Experimental): Topiramate 200 mg daily plus Aripiprazole 7.5mg daily
  Interventions: Drug: Topiramate 200, Aripiprazole 7.5mg

INTERVENTIONS:
Drug: Double Placebo — 1 capsule daily
  Arms: Double Placebo
Drug: Aripiprazole 15, placebo — 15 mg Aripiprazole daily plus placebo daily
  Other Names: Abilify, Topamax
  Arms: Aripiprazole 15, Placebo
Drug: Aripiprazole 7.5, Placebo — Aripiprazole 7.5 mg daily plus Placebo daily
  Arms: Aripiprazole 7.5, Placebo
Drug: Topiramate 100, Placebo — Topiramate 100 mg daily plus Placebo daily
  Arms: Topiramate 100mg, Placebo
Drug: Topiramate 200, Placebo — Topiramate 200 mg daily plus Placebo daily
  Arms: Topiramate 200, Placebo
Drug: Topiramate 100, Aripiprazole 15 — Topiramate 100 mg daily plus Aripiprazole 15mg daily
  Other Names: Abilify, Topamax
  Arms: Topiramate 100, Aripiprazole 5
Drug: Topiramate 100, Aripiprazole 7.5 — Topiramate 100 mg daily plus Aripiprazole 7.5mg daily
  Arms: Topiramate 100, Aripiprazole 7.5
Drug: Topiramate 100, Aripiprazole 15mg — Topiramate 100 mg daily plus Aripiprazole 15mg daily
  Other Names: Abilify; Topamax
  Arms: Topiramate 100, Aripiprazole 5
Drug: Topiramate 200, Aripiprazole 7.5mg — Topiramate 200 mg daily plus Aripiprazole 7.5mg daily
  Other Names: Abilify; Topamax
  Arms: Topiramate 200, Aripiprazole 7.5mg
Drug: Topiramate 200, Aripiprazole 15 — Topiramate 200mg daily plus Aripiprazole 15mg daily
  Other Names: Abilify; Topamax
  Arms: Topiramate 200, Aripiprazole 15

SUMMARY:
The current study investigates the effects of two potential alcohol treatment medications on drinking in a laboratory setting. Aripiprazole (APZ), effects dopamine and serotonin receptors with fewer limiting side effects seen with other atypical antipsychotics. Topiramate (TPMT), an antiepileptic, affects glutamate and GABA-A receptors and shows promise in reducing heavy drinking. Few studies have used two medications with such a diverse combination of actions to examine a potential synergistic effect on reducing alcohol consumption.

The primary aims are to:

1. determine if APZ and TPMT are each more effective than placebo, and the combination of APZ and TPMT is more effective than either drug alone or placebo, in reducing alcohol use in non-treatment seeking alcohol dependent subjects in a laboratory based alcohol self-administration experiment (ASAE)
2. examine a hypothesized dose-response for three doses of APZ (0, 7.5 mg/d and 15 mg/d) along with three doses of TPMT (0, 100mg/d and 200mg/d)
3. examine the putative mechanisms of action of APZ, TPMT alone and together on craving, subjective stimulation, candidate gene influences and other behavioral effects associated with alcohol consumption
4. establish the safety of giving APZ and TPMT together. Non-treatment seeking, alcohol dependent Participants (N=216) will be recruited from the community and randomly assigned to one of the 9 cells. Subjects drinking and safety is monitored over a 5-week titration to their target dose, leading to an in-laboratory alcohol self administration session, during which clinical and behavioral effects are assessed during access to alcohol. A 1 month follow-up assesses adverse events and drinking.

DETAILED DESCRIPTION:
Due to the modest effect of current pharmacotherapies, more effective treatments must be developed to optimally treat alcohol dependent patients. Treatments combining pharmacotherapies with different mechanisms of action may better address the diverse neurobiology of alcohol and the heterogeneity of alcoholics. However, little is known about how medication may affect behavior to reduce drinking. Aripiprazole (APZ), a partial dopamine agonist, affects dopamine and serotonin receptors without the limiting side effects seen with other atypical antipsychotics. Dopamine mediates reward based drinking and craving. Topiramate (TPMT), an antiepileptic, affects glutamate and GABA-A receptors and shows promise in reducing heavy drinking. Glutamate and GABA may mediate relief-based drinking and protracted withdrawal. Despite strong evidence that multiple neurotransmitters contribute to alcoholism, few studies have used two medications with such a diverse combination of actions to examine a potential synergistic effect on reducing alcohol consumption.

The present study will recruit 216 healthy, alcohol-dependent volunteers who are not currently seeking treatment for their alcohol dependence to learn more about how these medications may work.

The primary aims are to: (1) determine if APZ and TPMT are each more effective than placebo, and the combination of APZ and TPMT is more effective than either drug alone or placebo, in reducing alcohol use in non-treatment seeking alcohol dependent subjects in an alcohol self administration experiment (ASAE); (2) examine a hypothesized dose-response for three doses of APZ (0, 7.5mg/d and 15 mg/d) and three doses of TPMT (0, 100mg/d, 200mg/d); (3) examine the putative mechanisms of action of APZ, TPMT alone and together on craving, subjective stimulation, candidate gene influences and other behavioral effects associated with alcohol consumption; and (4) establish the safety of giving APZ and TPMT together. We will use of a 3 X 3 drug (7.5mg, 15mg APZ vs. placebo) by drug (100mg, 200mg TPMT vs. placebo) between-subjects factorial design. Participants are randomly assigned to one of 9 cells. Subjects drinking and safety is monitored over a 5-week titration to their target dose, leading to an in-laboratory alcohol self administration session, during which clinical and behavioral effects are assessed during access to alcohol. A 1 month follow-up assesses adverse events and drinking. The long term objectives of this research are to improve medications available for alcoholism treatment and inform research and theory on the mechanisms of action of such medications.

ELIGIBILITY:
Inclusion Criteria:

* must be non-treatment seeking for alcohol dependence
* a current DSM-IV-TR diagnosis of alcohol dependence supported by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders Patient Edition (SCID-I/P a minimum of ≥ 35drinks a week for men or ≥ 28 or more drinks a week for women
* must be suitable for outpatient treatment
* able to read English at an eighth grade level, understand their rights as provided by the informed consent, and be willing to sign an informed consent to participate in the study
* be between 21 and 65 years on age (inclusive)
* provide evidence of stable residence in the two months prior to enrollment and no plans to move for the next four months
* provide a verifiable contact person prior to randomization
* be in generally good health as determined by the physical exam, medical history, ECG and laboratory tests
* have a Body Mass Index >18kg/m2 and < 33 kg/m2
* if female, must be postmenopausal practicing an effective method of birth control, have negative pregnancy tests at randomization and before the ASAE;
* be willing to be adherent to medication dosing.

Exclusion Criteria:

* clinically significant medical abnormalities (i.e. ECG, hematological assessment, bilirubin > 150% of the upper limit of normal or ALT or AST elevations >300% the upper limit of normal, biochemistry including urinalysis, electrolytes,). (Persons with medical conditions that are adequately controlled by their primary care physician will not be excluded.)
* have significant alcohol withdrawal symptoms (clinical institute withdrawal assessment for alcohol revised (CIWA-Ar) >10
* a history of suicide; history of renal impairment or nephrolithiasis; creatinine clearance of <60 dl/minute
* pregnant or lactating or not using an adequate form of birth control
* taking other medications that may have an effect on alcohol consumption or are carbonic anhydrase inhibitors
* clinically significant diseases of the gastrointestinal system or active liver disease; subjects compelled to receive treatment to avoid imprisonment or loss of employment
* previously with a history of adverse reaction or hypersensitivity to either Topiramate or aripiprazole
* have a diagnosis of with schizophrenia or bipolar disorder and/or taking antipsychotics and other drugs that inhibit CYP3A4 or CYP2D6 isoenzymes
* history of seizures (e.g. epilepsy)
* patients currently diagnosed with a substance dependence diagnosis other than alcohol or tobacco
* patients who have participated in any clinical trial with an investigational agent within the past 30 days
* individuals with a reasonable expectation of being institutionalized during the course of the trial or pending legal charges
* pregnant or nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of alcoholic drinks consumed in a laboratory setting | 90 minutes
Safety and tolerability of the medications singly and in combination, compared to placebo | 4 years

SECONDARY OUTCOMES:
Drinks consumed during the medication titration period | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Swift, MD, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University Center for Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Haass-Koffler CL, Goodyear K, Zywiak WH, Leggio L, Kenna GA, Swift RM. Comparing and Combining Topiramate and Aripiprazole on Alcohol-Related Outcomes in a Human Laboratory Study. Alcohol Alcohol. 2018 May 1;53(3):268-276. doi: 10.1093/alcalc/agx108. PMID 29281033